CLINICAL TRIAL: NCT01224093
Title: A Multicentre, Observational, Prospective Study to Assess the Safety Profile of Rituximab in Combination With Chemotherapy in Patients With B Cell-lineage Chronic Lymphocytic Leukaemia (B-CLL)
Brief Title: An Observational Study on the Safety Profile of MabThera/Rituxan (Rituximab) in Combination With Chemotherapy in Patients With B Cell-lineage Chronic Lymphocytic Leukaemia (MABERYC)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25372
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Drug Therapy; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- First line
  Interventions: Drug: Chemotherapy; Drug: rituximab [MabThera/Rituxan]
- Relapsed/refractory
  Interventions: Drug: Chemotherapy; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: Chemotherapy — as prescribed
Drug: rituximab [MabThera/Rituxan] — as prescribed

SUMMARY:
This prospective observational study will evaluate the safety of MabThera/Rituxan (rituximab) in combination with chemotherapy in patients with previously untreated or relapsed/refractory B cell-lineage chronic lymphocytic leukaemia. Data will be collected from each patient for 6-12 months, depending on the prescribed chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* B cell-lineage chronic lymphocytic leukaemia (B-CLL)
* Prescribed with MabThera/Rituxan in combination with chemotherapy according to the approved SMPC
* Informed consent to data collection

Exclusion Criteria:

* Treatment with any marketed or non-marketed drug substance or experimental therapy within 4 weeks prior to first dose of study drug or participation in a clinical trial within 30 days prior to entering this study
* Any other tumour disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with B cell-lineage chronic lymphocytic leukaemia (B-CLL)
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety profile of MabThera/Rituxan in combination with chemotherapy in unselected CLL patients | 3 years

SECONDARY OUTCOMES:
Efficacy (Response rate, duration of response, progression-free survival) | 3 years
Chronic lymphocytic leukaemia (CLL) Comorboid Scale | 3 years
Quality-adjusted survival analysis (Q-TWIST methodology) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Spain (39):
  - Vitoria-Gasteiz, Alava
  - Alicante, Alicante
  - Elche, Alicante
  - Almería, Almeria
  - Palma de Mallorca, Balearic Islands
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Cadiz, Cadiz
  - Jerez de la Frontera, Cadiz
  - Puerto Real, Cadiz
  - Santander, Cantabria
  - Castellon, Castellon
  - Girona, Girona
  - Huelva, Huelva
  - Jaén, Jaen
  - Ferrol, La Coruña
  - Logroño, La Rioja
  - Las Palmas, Las Palmas
  - Las Palmas de Gran Canaria, Las Palmas
  - León, Leon
  - Lleida, Lerida
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Cartagena, Murcia
  - Lorca, Murcia
  - Pamplona, Navarre
  - Gijón, Principality of Asturias
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Tarragona, Tarragona
  - San Cristóbal de La Laguna, Tenerife
  - Santa Cruz de Tenerife, Tenerife
  - Alzira, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Bilbao, Vizcaya
  - Zaragoza, Zaragoza